CLINICAL TRIAL: NCT05250739
Title: Effect of Neuromuscular Training vs Strength Training in Chronic Ankle Instability
Brief Title: Neuromuscular Training vs Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DAVID CRUZ DÍAZ (Other)
Responsible Party: Sponsor-Investigator, DAVID CRUZ DÍAZ, Principal Investigator, University of Jaén
Organization: University of Jaén (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANKLEST
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent assessor blinded to the data collection was responsible for the allocation process. A list of the computer-generated number was employed to assign participants to experimental or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strength training (Experimental): Participants completed 16 training sessions of strength training during eight weeks.
  Interventions: Other: Strength training
- Neuromuscular training (Experimental): Participants completed 16 training sessions of neuromuscular training during eight weeks.
  Interventions: Other: Neuromuscular training
- Control group (No Intervention): The Control group received no intervention.

INTERVENTIONS:
Other: Strength training — Strength training was performed with resistance bands. The band was fastened to the unaffected ankle, while the participant was told to perform front and back pulls, as well as adduction and abduction movements with the affected ankle. They were told to control the ankle movement and to make it slow. Since the first day, they were told to perform the exercise pulling the band as if they wanted to make the resistance of 5 on a scale from 0 to 10.
  Arms: Strength training
Other: Neuromuscular training — consisted in a multi-station training with 6 exercises, increasing the difficulty progressively as the participants controlled the execution. The exercises were all performed barefoot and with the injured foot. These were a combination of standing and jumping exercises involving the injured ankle. The participants did not start the next progression until they perform a complete circuit in the level before.
  Arms: Neuromuscular training

SUMMARY:
Chronic ankle instability is a complex condition. Limited mobility, perceived instability, and recurrent ankle sprains are common characteristics that reduce the quality of life in subjects who suffer chronic ankle instability. Neuromuscular training and strength training has been recommended in chronic ankle instability management interventions. However, there are contradictory findings on results when comparing neuromuscular training, strength training, and control group.

DETAILED DESCRIPTION:
Participants were randomly assigned to the neuromuscular training group, strength training group, and control group with no intervention if participants met the inclusion criteria.

Neuromuscular training group. It consisted of a multi-station training with 6 exercises, increasing the difficulty progressively as the participants controlled the execution. The exercises were all performed barefoot and with the injured foot. These were a combination of standing and jumping exercises involving the injured ankle.

A strength training group was performed with resistance bands. The band was fastened to the unaffected ankle, while the participant was told to perform front and back pulls, as well as adduction and abduction movements with the affected ankle. Participants were told to control the ankle movement and to make it slow.

Control group received no intervention.

ELIGIBILITY:
Inclusion criteria were consistent with recommendations made from International Ankle Consortium16 and were checked before the intervention:

* To have suffered the first sprain at least 6 months before the beginning of the study.
* Cumberland ankle instability score ≤24.
* To be physically active.

Exclusion criteria.

* Participants could not have suffered an acute sprain in the 6 previous weeks to the beginning of the study.
* History of recent ankle surgery.
* Epilepsy or previous seizures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Self-reported instability | From baseline to eight weeks
  To determine the presence and severity of chronic ankle instability, participants completed the Cumberland Ankle Instability Tool, a valid and reliable instrument for measuring the severity of ankle instability. The Cumberland Ankle Instability Tool is a 9-item subjective questionnaire with a range score from 0 (severe instability) to 30 (normal stability)

SECONDARY OUTCOMES:
Ankle range of motion | From baseline to eight weeks
  Ankle dorsiflexion range of motion was assessed by the weight-bearing lunge test. The patient is positioned in a standing position facing a wall with the involved foot parallel with a tape measure which has been attached to the floor and the opposite leg placed behind in a tandem stance. A forward lunge is performed until the anterior knee tries to make contact with the wall with the heel firmly planted on the ground.
Dynamic balance | From baseline to eight weeks
  Dynamic balance has been measured by a simplified version of the Star Excursion Balance Test where the anterior, posteromedial and posterolateral reach directions were collected for statistical analysis.
Functional status | From baseline to eight weeks
  Function in daily living and sport activities were assessed by the Foot and Ankle Ability Measure. This questionnaire Is divided by two subscales of 21 items (daily living subscale) and 8 items (sports subscale). The obtained score is expressed as a percentage calculated by dividing the patient's score by max score and the lower percentage is related to the lower level of function.

CONTACTS AND LOCATIONS:
Overall Officials: David Cruz-Diaz, PhD, Principal Investigator — University of Jaen
Locations (1):
- University of Jaen, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No
Not allowed due to personal data legal protection issues.

REFERENCES:
- [Background] Halabchi F, Hassabi M. Acute ankle sprain in athletes: Clinical aspects and algorithmic approach. World J Orthop. 2020 Dec 18;11(12):534-558. doi: 10.5312/wjo.v11.i12.534. eCollection 2020 Dec 18. PMID 33362991
- [Background] Beynnon BD, Vacek PM, Murphy D, Alosa D, Paller D. First-time inversion ankle ligament trauma: the effects of sex, level of competition, and sport on the incidence of injury. Am J Sports Med. 2005 Oct;33(10):1485-91. doi: 10.1177/0363546505275490. Epub 2005 Jul 11. PMID 16009979
- [Background] Ahern L, Nicholson O, O'Sullivan D, McVeigh JG. Effect of Functional Rehabilitation on Performance of the Star Excursion Balance Test Among Recreational Athletes With Chronic Ankle Instability: A Systematic Review. Arch Rehabil Res Clin Transl. 2021 May 21;3(3):100133. doi: 10.1016/j.arrct.2021.100133. eCollection 2021 Sep. PMID 34589684